CLINICAL TRIAL: NCT01800201
Title: Automated Hovering to Improve Medication Adherence Among Myocardial Infarction Patients (Heartstrong)
Acronym: Heartstrong
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 817179; 1C1CMS331009-01-00 (Other Grant/Funding Number: Center for Medicare & Medicaid Innovation (CMMI))
Record Dates: First submitted 2013-02-25; First posted 2013-02-27 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Patients With Principal or Secondary Diagnosis Code of Intrntl Classification of Diseases, 9th Revision, (ICD-9-CM) 410 (Except When 5th Digit Was 2)
Keywords: Initial occurrence Acute Myocardial Infarction (AMI)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): The control group will have their claims data analyzed for a 12 month period. We will be examining these data for hospital admissions, new vascular events (AMI, stroke, acute coronary syndrome admission), or repeat or new cardiovascular procedures.
- Intervention (Experimental): The intervention group (1) will use GlowCaps, a remote monitoring and reminder pill bottle; (2) assigned an engagement advisor from the study team; (3) asked to provide study team with names and contact information of up to 3 family members or friends as support partners for med adherence. The study team will contact these people in order listed until 1 agrees to this role; (4) will select a 2-digit lucky number to be used as part of the sweepstakes-based engagement incentives in which eligibility to win will be conditional on med adherence; and (5) will determine preferences for Way to Health platform communication methods.The group receiving the program intervention will also have their claims data analyzed for the 12 months post-enrollment.
  Interventions: Behavioral: Electronic Pill Bottle, Incentives, Social Influence

INTERVENTIONS:
Behavioral: Electronic Pill Bottle, Incentives, Social Influence — The intervention group (1) will use GlowCaps, a remote monitoring and reminder pill bottle; (2) assigned an engagement advisor from the study team; (3) asked to provide study team with names and contact information of up to 3 family members or friends as support partners for med adherence. The study team will contact these people in order listed until 1 agrees to this role; (4) will select a 2-digit lucky number to be used as part of the sweepstakes-based engagement incentives in which eligibility to win will be conditional on med adherence; and (5) will determine preferences for Way to Health platform communication methods.The group receiving the program intervention will also have their claims data analyzed for the 12 months post-enrollment.
  Arms: Intervention

SUMMARY:
The goal of this proposal is to test the implementation of an innovative approach to improving health and lowering cost for a high risk population of patients with acute myocardial infarction (AMI) immediately post-hospitalization. The investigators will implement a new service delivery approach that will provide a foundation for a payment system that rewards keeping high-risk patients healthy and that deploys technology and a health care workforce of the future to implement prevention, care coordination, care process re-engineering, team-based care, and the use of data to support new care delivery models. This program is focused on coronary artery disease (CAD), but we expect that a successful implementation of this model will demonstrate a sustainable pathway to the three-part aim not just for CAD, but for many other conditions whose outcomes are highly sensitive to post-discharge coordination.

This proposal has three main principles:

1. Principles of behavioral economics that have been developed, refined, and tested over the past decade offer practical insights into health behaviors that were previously unavailable and are not reflected in existing care models.
2. New technology, typically wireless devices for pill bottles, and mobile telephones, make engagement with patients substantially easier and more immediate now than ever before.
3. While randomized clinical intervention trials provide exceptional confidence of comparative effectiveness in narrow interventions, they are slow and rigid and dont reflect the urgency that health care transformation currently requires. Principles of rapid cycle innovation are gaining acceptance as an alternative to or supplement of these traditional methods in supporting evidence for implementation success.

DETAILED DESCRIPTION:
The specific aims of this study are to:

1. Test the effectiveness of a state-of-the-art web-based portal with home-based wireless medication adherence devices and behavioral economic feedback mechanisms in preventing vascular events or re-hospitalization in the 12 months following hospital admission for AMI
2. Deploy a new model of evidence based evolutionary learning that uses rapid cycle innovation in 3 successive planning cycles over the 36 months of this proposal

Patients will be randomized into 1 of the 2 study groups.

1. The control group will have their health insurance claims records analyzed over a 12 month period for comparison to the participants in the intervention arm.
2. The intervention group:

(1) will use the GlowCaps, a remote monitoring and reminder pill bottle; (2) will be assigned an engagement advisor from the study team; (3) be asked to provide the study team with names and contact information of up to 3 family members or friends as support partners for medication adherence; (4) will be eligible for daily sweepstakes-based engagement incentives in which eligibility to win will be conditional on medication adherence; (5) can choose to modify their preferences for Way to Health platform communication methods during the study.

The group receiving the program intervention will also have their claims data analyzed for the 12 months post-enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to hospitals throughout New Jersey or at the University of Pennsylvania Health System who are discharged (or scheduled to be discharged) to their homes with a principal or secondary diagnosis code of International Classification of Diseases, 9th Revision, Clinical Modification (ICD-9-CM) 410 (except when the fifth digit was 2)
* a length of stay of 1 to 180 days
* Aged 18 to 80 years
* Be discharged to home
* Prescribed at least 2 of these 4 medication categories (statin, aspirin, beta-blocker, anti-platelet)

Exclusion Criteria:

* cannot give consent
* have a markedly shortened life expectancy (diagnosis of metastatic cancer, end-stage renal disease on dialysis, or dementia)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1509 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin GM Volpp, MD, PhD, Principal Investigator — University of Pennsylvania; David A Asch, MD, MBA, AB, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Volpp KG, Troxel AB, Mehta SJ, Norton L, Zhu J, Lim R, Wang W, Marcus N, Terwiesch C, Caldarella K, Levin T, Relish M, Negin N, Smith-McLallen A, Snyder R, Spettell CM, Drachman B, Kolansky D, Asch DA. Effect of Electronic Reminders, Financial Incentives, and Social Support on Outcomes After Myocardial Infarction: The HeartStrong Randomized Clinical Trial. JAMA Intern Med. 2017 Aug 1;177(8):1093-1101. doi: 10.1001/jamainternmed.2017.2449. PMID 28654972

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by University of Pennsylvania research staff from March 2013 through January 2015 and followed for one year.
Pre-assignment Details: No enrolled participants were excluded from the study before arm assignment
Groups:
- Intervention: The intervention group (1) will use the GlowCaps, a remote monitoring and reminder pill bottle; (2) will be assigned an engagement advisor from the study team; (3) asked to provide the study team with names and contact information of up to 3 family members or friends as support partners for medication adherence. The study team will contact these people in order listed until 1 agrees to serve in this role; (4) will select a 2-digit lucky number to be used as part of the sweepstakes-based engagement incentives in which eligibility to win will be conditional on medication adherence; and (5) will determine their preferences for Way to Health platform communication methods during the study.
  The group receiving the program intervention will also have their claims data analyzed for the 12 months post-enrollment.
Period: Overall Study
Arm/Group | Control | Intervention
Started | 506 | 1003
Completed | 503 | 1000
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — patient privacy concerns | 1 | 1
Not completed — did not want to use device | 0 | 1
Not completed — PI withdrawal, cognitive concerns | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 503 | 1000 | 1503
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 332 | 601 | 933
  >=65 years | 171 | 399 | 570
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (10.2) | 61.2 (10.4) | 61.0 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190 | 343 | 533
  Male | 313 | 657 | 970
Region of Enrollment [Number; unit: participants]
  United States | 503 | 1000 | 1503

OUTCOME MEASURES:

1. Primary Outcome: 1 -Year Survival Probability Rate: Vascular Readmissions or Death
Description: Primary outcome variable(s): 1- year survival probability rate for vascular inpatient readmission or death
Time Frame: Date of enrollment + 12 months
Measure: Number; unit: proportion of participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 503 | 1000
proportion of participants | .91 | .91

2. Secondary Outcome: 1 Year Survival Probability Rate All Cause Readmissions
Description: 1 year survival probability rate for all cause readmissions
Time Frame: Date of enrollment + 12 months
Measure: Number; unit: proportion of participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 503 | 1000
proportion of participants | .65 | .69

3. Secondary Outcome: Total Vascular Inpatient Readmissions
Description: This is the number of vascular inpatient admission events control vs. intervention
Time Frame: Date of enrollment + 12 months
Measure: Number; unit: readmissions
Arm/Group | Control | Intervention
Number analyzed (Participants) | 503 | 1000
readmissions | 62 | 119

4. Secondary Outcome: Proportion of Days Covered (PDC) for a Subset of Patients for Whom we Have Prescription Information
Description: Calculated by the proportion of days in which a patient has an active medication for all three medications (statin, beta blocker and antiplatelet). It is not the weighted average of the individual medication. This reflects the "intermediate" definition of adherence: our intermediate definition assumed that patients had been prescribed a medication for the entire study period if they ever filled that medication after discharge
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: PDC, mean
Arm/Group | Control | Intervention
Number analyzed (Participants) | 246 | 516
PDC, mean | .58 (0.35) | .61 (0.33)

ADVERSE EVENTS:
Time Frame: 1509 participants were enrolled starting in March 2013 through January 2015 and observed for one year. 6 patients withdrew. Adverse event data was collected for 1503 participants during all 12 months of their participation.
Description: We only have a report of deaths from medical claims if the patient died in the hospital, as a result we did not report on deaths in our manuscript due to incomplete data.
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 4/503 | 8/1000
Serious Adverse Events (participants affected / at risk) | 37/503 | 66/1000
Other Adverse Events (participants affected / at risk) | 0/503 | 0/1000
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=503) | Intervention (N=1000)
Intracranial Hemmorhage (Cardiac disorders) | 0 (0) | 5 (7) — intracranial hemorrhage as identified by ICD-9: 430, 431,432.0, 432.9, 853, 430, 431
Liver Failure (Renal and urinary disorders) | 1 (1) | 1 (1) — Liver Failure as defined by ICD-9: 570.0, 573.3
Heart Block (Cardiac disorders) | 1 (1) | 4 (6) — Heart Block as defined by following ICD-9: 426.9, 426.0, 426.12, 426.13
Rhabdomyolysis (Renal and urinary disorders) | 1 (1) | 4 (4) — Rhabdomyolysis as defined by ICD-9: 728.88, 791.2, 791.3
GI Hemmorhage/Ulcer (Gastrointestinal disorders) | 12 (16) | 12 (14) — GI Hemmorhage/Ulcer as identified by ICD-9: 578.0, 578.1, 578.9, 569.3, 531, 532, 533, 534:
Syncope (Blood and lymphatic system disorders) | 6 (6) | 13 (16) — Synope as identifed by ICD-9: 780.2
Bradycardia (Cardiac disorders) | 14 (15) | 27 (29) — Bradycardia as identified by ICD-9: 427.89
Unspecified Hemmorhage (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — Unspecified Hemmorhage as identified as ICD-9: 459.0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No